CLINICAL TRIAL: NCT02631408
Title: Application of Intrawound Vancomycin Powder to Reduce Surgical Site Infections in Spinal Fusion Surgery - A Prospective, Randomized, Controlled Trial
Brief Title: Intrawound Vancomycin Powder in Spinal Fusion Surgery
Acronym: iVRCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orthopedic Hospital Vienna Speising (Other)
Responsible Party: Principal Investigator, Lukas Panzenboeck, Dr. Lukas Panzenboeck, Orthopedic Hospital Vienna Speising
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: iVRCT1_4
Record Dates: First submitted 2015-12-12; First posted 2015-12-16 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Spinal Fusion Acquired
Keywords: spinal fusion; topical antibiotics; vancomycin; surgical site infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Vancomycin; Powders; Solutions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): No additional treatment. Routine iv. antibiotic prophylaxis only.
- Vancomycin Group (Experimental): Vancomycin powder is applied before wound closure. Routine iv. prophylaxis stays unchanged
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Locally, intrawound applied vancomycin powder
  Other Names: Vancomycin Hydrochloride, Powder for Solution for Infusion
  Arms: Vancomycin Group

SUMMARY:
Vancomycin powder (for solution for Infusion) will be investigated (off-label usage) in spinal fusion surgery. The powder will be locally administered into to the wound cavity before wound closure.

Hypothesis: Locally applied vancomycin powder leads to a reduction in postoperative surgical site infections

DETAILED DESCRIPTION:
Vancomycin is being widely used as an antibiotic agent for intravenous and topical use. The surgical application of vancomycin powder in Austria is limited as there is no powder with marketing authorization for intraoperative, intrawound usage. Previous reports widely document the application of vancomycin powder for solution for infusion. The powder is not soluted, but instead directly spread throughout the wound surface. Limited data is available for spinal fusion surgery, mostly retrospective studies. Results were promising, but the low evidence level does not allow for a conclusion regarding routine usage. Additional randomized, controlled trials are necessary to further investigate this matter.

This trial aims to investigate Vancomycin powder "Xellia" 1000mg, which has a Marketing authorization, in an off-label usage (intrawound, intraoperatively) in spinal fusion surgery. The investigational medicinal product will be used unmodified.

ELIGIBILITY:
Inclusion Criteria:

* Planned TLIF (transforaminal lumbar interbody fusion) or PLIF (posterolateral lumbar interbody fusion) surgery
* TLIF/PLIF fusion length of one or two motion-segments OR
* One motion-segment TLIF/PLIF in conjunction with one motion-segment decompression surgery or microscopic disc surgery (microdiscectomy)
* Fusions within L1 (first lumbar vertebra) through S1 (sacrum)
* Age of 18-years or older
* Signed informed consent

Exclusion Criteria:

* Preoperative inflammatory or infectious state (C-reactive protein levels above 10mg/l)
* Allergic to vancomycin, teicoplanin or penicillin
* Preexisting auto-immune disease with an impaired immune system
* Current post-traumatic vertebral injury (e.g. vertebral split fracture)
* Preexisting Renal impairment
* Preexisting cochlea damage
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2015-08; Primary Completion 2019-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
SSI rate | 1 year
  Rate of superficial and deep surgical site infections (according to CDC criteria)

SECONDARY OUTCOMES:
C-reactive protein | 7 days
  Course of postoperative CRP levels
Revision rate | 1 year
  Revision rate due to surgical site infections

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Becker, MD, Principal Investigator — Orthopedic Hospital Speising; Lukas Panzenboeck, MD, Study Chair — Orthopedic Hospital Speising
Locations (1):
- Orhopedic Hospital Speising, Vienna, Austria